CLINICAL TRIAL: NCT03778398
Title: The Effect Of Music Therapy On Upper Extremity Functions In Adolescents With Cerebral Palsy
Brief Title: Music Therapy In Adolescents With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMU FTR
Record Dates: First submitted 2018-12-02; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Palsy
Keywords: music therapy; cerebral palsy; piano training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurologic music therapy (Experimental): Patients will receive 2 days of 40 minutes per week, total 3 months of customized piano training. Each session will be started with finger warming exercises, then with the right hand, left handed and with both hands, a simple pentatonic array will be played. In the following lessons, notes will be marked with colors and simple songs will be taught.
  Interventions: Other: Neurologic music therapy

INTERVENTIONS:
Other: Neurologic music therapy — Customized piano training

SUMMARY:
Purpose of the study;

* To improve the upper extremity motor functions of patients with adolescent cerebral palsy,
* Prevent treatment interruptions as age progresses,
* Increase the hand functions of children with cerebral palsy and to increase their living standards.

Hand functions will be assessed with MACS (Manual Ability Classification System), hand dynamometer, box-block test, 9 hole peg test, pressing velocity measured with Cubase MIDI (musical instrument data interface) program. Patients will receive 2 days of 40 minutes per week, total 3 months of customized piano training. Each session will be started with finger warming exercises, then with the right hand, left handed and with both hands, a simple pentatonic array will be played. In the following lessons, notes will be marked with colors and simple songs will be taught. At the end of 3 months, the tests will be repeated.

DETAILED DESCRIPTION:
Cerebral palsy is the development, movement and posture disorder that causes the limitation of activity which is thought to be caused by non-progressive disorders in the fetal or infant brain. Intensive rehabilitation program begins in early childhood; However, adults with cerebral palsy are less likely to receive rehabilitative interventions. There is a great need for effective upper extremity rehabilitation studies that motivate the patient in CP (cerebral palsy) rehabilitation after childhood. Therapeutic Instrumental Music Performance (TIMP) is one of the three techniques of neurological music therapy techniques for motor rehabilitation. This technique uses instruments to strengthen functional motor patterns. There are very few studies on TIMP in individuals with cerebral palsy and these studies have not been performed on patients with adolescent cerebral palsy.

Purpose of the study;

* To improve the upper extremity motor functions of patients with adolescent cerebral palsy,
* Prevent treatment interruptions as age progresses,
* Increase the hand functions of children with cerebral palsy and to increase their living standards.

Inclusion Criteria:

* Being 11-18 years old
* To be diagnosed with cerebral palsy
* Not have been previously trained piano
* To have enough cognitive function to perform commands
* Accepted to participate in the study

Criteria for not being included in research:

* Having cognitive disorder
* Advanced visual impairment, visual field defect
* To be previously trained for piano
* Another disease preventing upper extremity movements

Hand functions will be assessed with MACS (Manual Ability Classification System), hand dynamometer, box-block test, 9 hole peg test, pressing velocity measured with Cubase MIDI (musical instrument data interface) program. Patients will receive 2 days of 40 minutes per week, total 3 months of customized piano training. Each session will be started with finger warming exercises, then with the right hand, left handed and with both hands, a simple pentatonic array will be played. In the following lessons, notes will be marked with colors and simple songs will be taught. At the end of 3 months, the tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Being 11-18 years old
* To be diagnosed with cerebral palsy
* Not have been previously trained piano
* To have enough cognitive function to perform commands
* Accepted to participate in the study

Exclusion Criteria:

* Having cognitive disorder
* Advanced visual impairment, visual field defect
* To be previously trained for piano
* Another disease preventing upper extremity movements

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Improved hand function | 3 months
  Improvement on MACS (Manual Ability Classification System)
Improved hand strength | 3 months
  Improvement on hand dynamometer and pressing velocities measured by Cubase MIDI (musical instrument data interface) program
Improved fine motor skills | 3 months
  Improvement on box-block test
Improved fine motor skills | 3 months
  Improvement on 9 hole peg test

SECONDARY OUTCOMES:
Improved hand coordination | 3 months
  observational, development of the ability to play the piano with two hands

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No